CLINICAL TRIAL: NCT07082569
Title: Effect of Ventilation Mode in the Pupillary Light Reflex: A Crossover Study
Acronym: EYE-BREATH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Evangelismos Hospital (Other)
Responsible Party: Principal Investigator, Charikleia Vrettou, Principal Investigator, Evangelismos Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: PSVCPC
Record Dates: First submitted 2025-07-05; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Mechanical Ventilation; Critical Illness
Keywords: Critical illness; Mechanical ventilation; Pupillary light reflex; Automated pupillometry; Neurological Pupil Index
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Each participant will receive three different modes of mechanical ventilation (Volume Control, Pressure Control, Pressure-Regulated Volume Control) in a randomized order. Pupillometry measurements will be taken after each mode, with a 15-minute washout period between modes.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be masked to the ventilation mode sequence applied during each pupillometry measurement. Pupillometry data will be anonymized and coded prior to statistical analysis to prevent bias in outcome evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence A: VC → PC → PRVC (Experimental): Participants receive mechanical ventilation in the following sequence: Volume Control (VC), followed by Pressure Control (PC), then Pressure-Regulated Volume Control (PRVC). Pupillometry is performed after each mode following a 15-minute stabilization period.
  Interventions: Other: Volume Control Ventilation; Other: Pressure Control Ventilation; Other: Pressure-Regulated Volume Control (PRVC)
- Sequence B: VC → PRVC → PC (Other): Participants receive mechanical ventilation in the following sequence: Volume Control (VC), followed by Pressure-Regulated Volume Control (PRVC), then Pressure Control (PC). Pupillometry is performed after each mode following a 15-minute stabilization period.
  Interventions: Other: Volume Control Ventilation; Other: Pressure Control Ventilation; Other: Pressure-Regulated Volume Control (PRVC)
- Sequence C: PC → VC → PRVC (Other): Participants receive mechanical ventilation in the following sequence: Pressure Control (PC), followed by Volume Control (VC), then Pressure-Regulated Volume Control (PRVC). Pupillometry is performed after each mode following a 15-minute stabilization period.
  Interventions: Other: Volume Control Ventilation; Other: Pressure Control Ventilation; Other: Pressure-Regulated Volume Control (PRVC)
- Sequence D: PC → PRVC → VC (Other): Participants receive mechanical ventilation in the following sequence: Pressure Control (PC), followed by Pressure-Regulated Volume Control (PRVC), then Volume Control (VC). Pupillometry is performed after each mode following a 15-minute stabilization period.
  Interventions: Other: Volume Control Ventilation; Other: Pressure Control Ventilation; Other: Pressure-Regulated Volume Control (PRVC)
- Sequence E: PRVC → VC → PC (Other): Participants receive mechanical ventilation in the following sequence: Pressure-Regulated Volume Control (PRVC), followed by Volume Control (VC), then Pressure Control (PC). Pupillometry is performed after each mode following a 15-minute stabilization period.
  Interventions: Other: Volume Control Ventilation; Other: Pressure Control Ventilation; Other: Pressure-Regulated Volume Control (PRVC)
- Sequence F: PRVC → PC → VC (Other): Participants receive mechanical ventilation in the following sequence: Pressure-Regulated Volume Control (PRVC), followed by Pressure Control (PC), then Volume Control (VC). Pupillometry is performed after each mode following a 15-minute stabilization period.
  Interventions: Other: Volume Control Ventilation; Other: Pressure Control Ventilation; Other: Pressure-Regulated Volume Control (PRVC)

INTERVENTIONS:
Other: Volume Control Ventilation — Standard mode of mechanical ventilation delivering a preset tidal volume. Commonly used in ICU patients requiring controlled ventilation.
Other: Pressure Control Ventilation — Pressure-targeted ventilation mode that delivers breaths at a fixed pressure. Commonly used in critically ill patients.
Other: Pressure-Regulated Volume Control (PRVC) — Hybrid ventilation mode that automatically adjusts inspiratory pressure to achieve a preset tidal volume.

SUMMARY:
The goal of this clinical trial is to explore whether different modes of mechanical ventilation affect pupillary constriction velocities in critically ill patients without brain injury. The study aims to determine whether the type of mechanical ventilation (volume control, pressure control, or pressure-regulated volume control) influences the maximum and mean constriction velocity measured by automated pupillometry. The trial also investigates whether changes in pupil dynamics reflect subtle alterations in brainstem-autonomic interaction induced by ventilation mode.

The comparison involves volume control, pressure control, and pressure-regulated volume control in a randomized crossover design to assess whether ventilation mode has a measurable effect on pupil response.

Eligible participants will be intubated ICU patients receiving assist control ventilation who are not yet ready for spontaneous breathing trials. Serial pupillometry measurements will be conducted while participants are ventilated with each mode for at least 15 minutes. Sedation and lighting conditions will remain consistent throughout the protocol. Participants with acute or chronic neurologic conditions or ventilator dyssynchrony will be excluded.

DETAILED DESCRIPTION:
This is a prospective, randomized, crossover study designed to evaluate the effect of different modes of mechanical ventilation on pupillary constriction velocity in critically ill patients. Recent data suggest that even in the absence of direct pulmonary or neurologic injury, mechanical ventilation with positive pressure may impact brain function, possibly through vagal-brainstem-autonomic pathways. These effects may be subtle and difficult to detect with standard neurological examination but may be reflected in changes in the dynamic pupillary light reflex.

The pupillary light reflex (PLR), measured using automated infrared pupillometry, provides a quantitative, non-invasive assessment of brainstem and autonomic nervous system function. IThe investigators aim to determine whether the PLR, specifically, the mean and maximum constriction velocity, differs across three commonly used ventilation modes: Volume Control (VC), Pressure Control (PC), and Pressure-Regulated Volume Control (PRVC).

All included participants will be mechanically ventilated, sedated, and not yet candidates for spontaneous breathing trials. Exclusion criteria include any acute or chronic neurologic disorder or signs of ventilator dyssynchrony. Sedation regimens (e.g., propofol, remifentanil, dexmedetomidine) will be kept constant during the study, and ambient light will remain unchanged.

Each participant will undergo the three ventilation modes in a randomized order, with each mode applied for a minimum of 15 minutes to ensure washout before pupillometry measurements are performed. Physiological parameters such as respiratory rate, minute ventilation, FiO₂, heart rate, and mean arterial pressure will be recorded in parallel with pupil measurements. Blood gas analysis and full pupillometry data, including pupil size, constriction and dilation velocities, latency, and the Neurological Pupil Index (NPi), will also be collected.

The primary outcome is the difference in maximum pupillary constriction velocity between ventilation modes. Secondary outcomes include mean constriction velocity, NPi, and other pupillary metrics. Based on pilot data, a total of 36 participants are required to detect a significant difference in the primary outcome. Statistical analysis will include repeated measures ANOVA or the Friedman test, with post hoc Wilcoxon Signed-Rank testing as appropriate.

The findings of this study may provide support for the use of pupillometry as a tool to assess subtle CNS effects of mechanical ventilation and could support the theory of ventilation-brainstem interactions during mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria

* Adult patients (≥18 years old)
* Receiving positive-pressure mechanical ventilation
* Under light or no sedation (e.g., RASS score between -2 and 0)
* Clinically assessed by the treating physician as not yet ready for weaning from mechanical ventilation
* Hemodynamically stable at the time of measurement
* Presence of an arterial catheter in place for blood gas analysis
* Written informed consent obtained from the patient's legal representative Exclusion Criteria
* Acute or chronic neurological disease affecting brainstem function or pupillary responses
* Dyssynchrony with the ventilator or need for high ventilatory support adjustments
* Facial injuries, edema, or conditions precluding accurate pupillometry
* Use of neuromuscular blocking agents within the prior 6 hours
* Severe metabolic or acid-base imbalances that may influence autonomic regulation
* Concurrent participation in another interventional study that could affect neurological or autonomic outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Pupillary Constriction Velocity | At 30 minutes after each ventilation mode initiation (VC, PC, PRVC).
  Change in maximum pupillary constriction velocity (mm/s) in response to standardized light stimulus, as measured by the NPi-200 pupillometer, under three modes of mechanical ventilation: Volume Control (VC), Pressure Control (PC), and Pressure-Regulated Volume Control (PRVC).

SECONDARY OUTCOMES:
Neurological Pupil Index (NPi) | At 30 minutes after each ventilation mode initiation (VC, PC, PRVC).
  Change in NPi value recorded under each ventilation mode, reflecting pupillary reactivity and brainstem function.
Constriction Latency | At 30 minutes after each ventilation mode initiation (VC, PC, PRVC).
  Change in latency to onset of pupil constriction (seconds), measured using the NPi-200.
Dilation Velocity | At 30 minutes after each ventilation mode initiation (VC, PC, PRVC).
  Change in maximum dilation velocity (mm/s) following light stimulus, measured with the NPi-200.
Maximum Pupil Diameter | At 30 minutes after each ventilation mode initiation (VC, PC, PRVC).
  Change in maximum pupil diameter (mm) measured before light stimulation under each ventilation mode.
Minimum Pupil Diameter | At 30 minutes after each ventilation mode initiation (VC, PC, PRVC).
  Change in minimum pupil diameter (mm) recorded after light stimulation.
Percent Constriction | At 30 minutes after each ventilation mode initiation (VC, PC, PRVC).
  Percent change in pupil diameter from baseline in response to light stimulus.

OTHER OUTCOMES:
Exploratory Outcome Measure - Heart Rate Variability (HRV) | Time interval between 15-30 minutes after the initiation of each ventilation mode (VC, PC, PRVC)
  HRV derived from ECG to explore autonomic nervous system modulation across ventilation modes (optional, if data acquisition becomes feasible).
Systolic Blood Pressure (mmHg) | At 30 minutes after each ventilation mode initiation (VC, PC, PRVC).
  Systolic blood pressure will be recorded during each ventilation mode to assess cardiovascular stability.
Diastolic Blood Pressure (mmHg) | At 30 minutes after each ventilation mode initiation (VC, PC, PRVC).
  Diastolic blood pressure will be recorded during each ventilation mode to assess cardiovascular stability.
Mean Arterial Pressure (mmHg) | At 30 minutes after each ventilation mode initiation (VC, PC, PRVC).
  Mean arterial pressure (MAP) will be recorded to evaluate overall hemodynamic stability.
Heart Rate (beats per minute) | At 30 minutes after each ventilation mode initiation (VC, PC, PRVC).
  Heart rate will be recorded to evaluate cardiovascular stability.
Arterial Partial Pressure of Oxygen, PaO₂ (mmHg) | At 30 minutes after each ventilation mode initiation (VC, PC, PRVC).
  PaO₂ will be measured via arterial blood gas to assess oxygenation.
Arterial Partial Pressure of Carbon Dioxide, PaCO₂ (mmHg) | At 30 minutes after each ventilation mode initiation (VC, PC, PRVC).
  PaCO₂ will be measured via arterial blood gas to assess ventilation efficiency.
Tidal Volume (mL) | At 30 minutes after each ventilation mode initiation (VC, PC, PRVC).
  Tidal volume will be recorded to ensure ventilator setting consistency.
Respiratory Rate (breaths per minute) | At 30 minutes after each ventilation mode initiation (VC, PC, PRVC).
  Respiratory rate will be recorded to monitor respiratory drive and ventilation stability.
Minute ventilation (L/min) | At 30 minutes after each ventilation mode initiation (VC, PC, PRVC).
  Minute ventilation will be recorded to assess ventilatory effectiveness and ensure consistency across modes.
Ambient Illumination (lux) | At 30 minutes after each ventilation mode initiation (VC, PC, PRVC).
  Ambient light intensity will be recorded to confirm consistent lighting conditions for pupillometry.

CONTACTS AND LOCATIONS:
Overall Officials: Charikleia S Vrettou, MD, PhD, Principal Investigator — !st ICU dpt., Evangelismos General Hospital
Locations (1):
- !st ICU dpt., Evangelismos Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to primary and secondary outcome measures will be made available to other researchers upon reasonable request, after publication of the main study results.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months after publication of the primary manuscript and continuing for 3 years.
Access Criteria: Access will be granted to qualified researchers for scientifically sound proposals. Requesters will need to submit a brief proposal outlining the purpose and methods of the secondary analysis.
URL: https://www.evaggelismos-hosp.gr/index.php/2016-08-29-13-40-56/org-dieuthunsh-iatrikhs-yphresias/org-diu-b-pathologikos-tomeas/pan-kliniki-entatikis

REFERENCES:
- [Background] Sibbald B, Roberts C. Understanding controlled trials. Crossover trials. BMJ. 1998 Jun 6;316(7146):1719. doi: 10.1136/bmj.316.7146.1719. No abstract available. PMID 9614025
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Muppidi S, Adams-Huet B, Tajzoy E, Scribner M, Blazek P, Spaeth EB, Frohman E, Davis S, Vernino S. Dynamic pupillometry as an autonomic testing tool. Clin Auton Res. 2013 Dec;23(6):297-303. doi: 10.1007/s10286-013-0209-7. Epub 2013 Jul 24. PMID 23880969
- [Background] Bassi TG, Rohrs EC, Fernandez KC, Ornowska M, Nicholas M, Gani M, Evans D, Reynolds SC. Transvenous Diaphragm Neurostimulation Mitigates Ventilation-associated Brain Injury. Am J Respir Crit Care Med. 2021 Dec 15;204(12):1391-1402. doi: 10.1164/rccm.202101-0076OC. PMID 34491883
- [Background] Cinnella G, Conti G, Lofaso F, Lorino H, Harf A, Lemaire F, Brochard L. Effects of assisted ventilation on the work of breathing: volume-controlled versus pressure-controlled ventilation. Am J Respir Crit Care Med. 1996 Mar;153(3):1025-33. doi: 10.1164/ajrccm.153.3.8630541.
- [Background] Walter K. Mechanical Ventilation. JAMA. 2021 Oct 12;326(14):1452. doi: 10.1001/jama.2021.13084. No abstract available. PMID 34636861